CLINICAL TRIAL: NCT02770989
Title: A Clinical Trial for the Assessment of the Safety and Performance of the Vimecon Laser Cardiac Ablation Instrument (CAI) for the Interventional Treatment of Paroxysmal Atrial Fibrillation (AF)
Brief Title: Vimecon CAI Trial for the Interventional Treatment of Paroxysmal Atrial Fibrillation (AF)
Acronym: CAI
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Design change
Sponsor: Vimecon GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VMC-001
Record Dates: First submitted 2015-12-10; First posted 2016-05-12 (Estimated); Last update posted 2018-12-13 (Actual); Status verified 2018-10

CONDITIONS: Atrial Fibrillation
Keywords: Cardiac Ablation; Safety; Performance; Laser
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vimecon Laser CAI Cardiac Ablation (Experimental): Ablation of the cardiac tissue by the use of the Vimecon Laser CAI (Cardiac Ablation Instrument).
  Interventions: Procedure: Vimecon Laser CAI percutaneous cardiac ablation

INTERVENTIONS:
Procedure: Vimecon Laser CAI percutaneous cardiac ablation — The Vimecon Laser CAI catheter is entered through the femoral vein to access the pulmonary vein (PV) area in the heart in order to ablate the cardiac wall near the PV to create scar tissue and to isolate the PV in order to treat atrial fibrillation.

SUMMARY:
This study is a prospective, non-randomized, single arm, multicenter, CE marking trial for patients with paroxysmal atrial fibrillation to undergo an ablation of the cardiac tissue near the PV.

DETAILED DESCRIPTION:
The objective of this clinical investigation is to confirm the safety and performance of the Vimecon® Laser Cardiac Ablation Instrument when creating scar tissue within the cardiac wall for the treatment of atrial fibrillation.

Up to 66 patients with paroxysmal atrial fibrillation refractory to at least one antiarrhythmic medications (Class I or III) are enrolled. with an expected 10% dropout; 59 per protocol patients are required.

The study duration will be 18 month with a 6 month enrollment period and 12 month follow-up. Interim follow-up visits are at post procedure, 1 Month, 3 Months, 6 Months and 12 Months.

The baseline and follow up tests are standard of care. Additional optional tests are an esophageal endoscopy for determination of potential fistula formation and a cerebral MRI for micro embolism post treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 to 75 years.
2. Patients with intention to be treated for paroxysmal atrial fibrillation. AND unresponsive to ≥1 antiarrhythmic drug (class I or III) AND at least 2 episodes in the last 12 months, 1 of them documented.
3. Patient should be on an anticoagulation therapy according to the international guidelines (per ACC/AHA//ESC Practice Guidelines)
4. Left atrial (LA) size < 50 mm
5. Symptomatic AF (EHRA-Score ≥ 2)
6. Accessibility of femoral vein and pulmonary veins
7. All patients willing to comply with the study protocol for at least 12 months

Exclusion Criteria:

1. 1. Inability to give written informed consent
2. NYHA Class III and IV
3. Hyperthyroidism
4. Reversible causes of the AF like Pericarditis, Electrolytic imbalance
5. Left Atrial Thrombus formation
6. Structural heart disease disturbing accessibility for AF ablation.
7. Valvular AF, permanent and long-standing persistent AF, currently present Atrial Flutter
8. Any valvular dysfunction more than II°
9. Systemic infections or endocarditis.
10. Impaired left ventricular function with an ejection fraction of less than 35%
11. Kidney dysfunction >Class III with a GFR of less than 35 mL per minute
12. TIA or stroke within the last 6 months
13. Pregnant and breastfeeding Women
14. Previous relevant cardiac surgery (e.g. ASD, PFO, Maze, AICD, pacemaker, congenital heart disorders or valve replacement).
15. Previous ablation of the pulmonary vein.
16. Known or suspected atrial myoma
17. Subject has co-morbid conditions that place the subject at an unacceptable risk (e.g., severe chronic obstructive pulmonary disease, hepatic failure, cerebral degenerative diseases, immunosuppressive abnormalities, hypercoagulable state, nervous system disease and hematological abnormalities.)
18. Contraindicated for the protocol defined anticoagulation plan (per ACC/AHA//ESC Practice Guidelines)
19. Patients with known allergic reactions to the local anesthetic, sedatives, x-ray dye, heparin, protamine, components of the catheter (platinum, iridium, stainless steel) or other agents administered during the procedure.
20. AV-Block IIº and IIIº
21. Contraindication for femoral vein and pulmonary veins access (e.g.: femoral Stent graft, excessive calcification, previous surgical interventions in or adjacent to the femoral veins that impede femoral access)
22. Contraindications for the transseptal approach (e.g.: previous inter-atrial septal patch or surgical interventions in or adjacent to the intro atrial septum)
23. MI in the last 3 months.
24. Enrolled in another clinical trial with a non-CE marked device which has not yet reached its primary endpoint

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2016-03; Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Safety assessment, free of any Major Adverse Events's or safety events within the first three (3) months after the treatment.. | < month-3
  Safety:
  • Evaluating the proportion of subjects free from experiencing Serious Adverse Events related to the catheter ablation procedure (Major Adverse Events's or safety events) within the first three (3) months after the treatment.
  Major adverse events (MAE, Safety events) associated with the catheter ablation procedure include:
  * Cardiac tamponade
  * Thromboembolic events including pulmonary embolism and stroke
  * Complete heart block
  * Acute myocardial infarction
  * Phrenic nerve palsy
  * Atrio-esophageal fistula
  * Vascular complications
  * Death

CONTACTS AND LOCATIONS:
Overall Officials: René Spaargaren, Dr., Study Director — Director Clinical Affairs
Locations (3):
- ZNA Middelheim, Antwerp, Belgium
- Na Homolce Hospital, Prague, Czechia
- "Herz- und Diabeteszentrum NRW Klinik für Kardiologie", Bad Oeynhausen, Germany

IPD SHARING:
Plan to Share IPD: No